CLINICAL TRIAL: NCT05823285
Title: A Phase 1 Study to Investigate the Safety, Tolerability，Pharmacokinetics, Immunogenicity and Preliminary Effectiveness of QLS31903 Injection in Subjects With Advanced Solid Tumors
Brief Title: A Study Evaluates the Safety, Pharmacokinetics, Immunogenicity and Efficacy of QLS31903 in Advanced Solid Tumor Patients
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Qilu Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: QLS31903-101
Record Dates: First submitted 2023-03-23; First posted 2023-04-21 (Actual); Last update posted 2023-04-21 (Actual); Status verified 2023-04

CONDITIONS: Advanced Solid Tumors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- QLS31903 (Experimental): 0.01μg/kg-2.16 μg/kg QLS31903 for injection
  Interventions: Drug: QLS31903

INTERVENTIONS:
Drug: QLS31903 — 0.01μg/kg-2.16 μg/kg QLS31903 for injection

SUMMARY:
The purpose of the study is to evaluate safety, pharmacokinetics,immunogenicity and efficacy of QLS31903 alone in the treatment of advanced cancer.

ELIGIBILITY:
Key Inclusion Criteria:

* 18 years or older, 40kg or heavier
* Histologically or cytologically confirmed diagnosis of advanced solid tumor （For phase 1b, patients must have solid tumor with GPC3+ )
* Standard treatment failed or standard treatment intolerant, no standard treatment
* Adequate hepatic, hematologic, and renal function

Key Exclusion Criteria:

* Anti-tumor treatment within 4 weeks prior to the first QLS31903 administration,except a few specific conditions
* Other clinical trial within 4 weeks prior to the first QLS31903 administration
* Receipt of a live or live attenuated vaccine within 30 days prior to the first QLS31903 administration
* Prior treatment targeted on GPC3
* HBsAg/HBcAb positive and HBV-DNA>10,000 copy/mL;HCV-Ab positive and HCV-RNA>1,000 copy/mL
* CNS metastasis (except asymptomatic brain metastases or symptomatic brain metastases after treatment stable for more than 4 weeks) and/or carcinomatous meningitis or leptomeningeal disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2023-03-22 (Actual); Primary Completion 2025-06-15 (Estimated); Study Completion 2027-06-15 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose（MTD）for Phase 1a | 21days or 14 days after the first target dose(whichever is longer）
  The MTD is determined by the number of the participants in cohort who suffer a dose-limiting toxicity (DLT). The MTD is defined as the former dose at which more than one third of the participants develop a DLT. If no DLTs are observed, the MTD is not reached.
Recommended phase 2 dose(RP2D) for Phase 1a | Duration of study, approximately 24 months
  The RP2D is defined as the dose level chosen by Safety Monitoring Committee(SMC)
Objective Response Rate (ORR) for phase 1b | From fist administration of QLS31903 to disease progression，death，loss to follow up,withdrawal of consent,initiation of a new anticancer therapy,study completion/closure,whichever came first, assessed up to 24 months
  ORR is the percentage of patients with best response of CR and PR

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoyan Kang, PhD, Study Chair — Qilu Pharmaceutical Co., Ltd.
Locations (1):
- Fudan Zhongshan Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No